CLINICAL TRIAL: NCT04336878
Title: Exploring the Feasibility and Acceptability of Integrating a Habit-based Intervention for Pregnant Women With Overweight or Obesity Into Existing Antenatal Care Pathways on the Island of Ireland: The HHIPBe Feasibility Study
Brief Title: Healthy Habits in Pregnancy and Beyond
Acronym: HHIPBe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: University of Leeds (Other); University College, London (Other); Belfast Health and Social Care Trust (Other); Western Health and Social Care Trust (Other); Sligo General Hospital (Other); Our Lady of Lourdes Hospital, Drogheda (Other Government)
Responsible Party: Principal Investigator, Michelle McKinley, Professor, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: QUB:B19/35 CHI/5434/2018; 266602 (Other: IRAS)
Record Dates: First submitted 2020-01-04; First posted 2020-04-07 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Overweight and Obesity; Pregnancy Related
Keywords: Gestational weight gain; Habit formation; Diet; Physical Activity; Behaviour change intervention
MeSH Terms: conditions — Overweight; Obesity; Gestational Weight Gain; Motor Activity | interventions — Pregnancy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the nature of the trial, it will not be possible to blind participants or intervention facilitators to group allocation. Researchers involved in collecting outcome data will not have access to details of group allocation and we will attempt to retain this blinding throughout. Participants will be asked not to discuss their group allocation with the researchers. Fidelity of blinding will be assessed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Habits in Pregnancy and Beyond intervention (Experimental): Intervention delivered in early pregnancy during an existing antenatal appointment. 1:1 intervention session (15-20 minutes) with the intervention facilitator (clinician/researcher). Participants provided with a self-guided leaflet for weight management focusing on making 10 simple diet and activity behaviours habitual, including advice on food choice & purchasing, portion size, eating behaviour & keeping active. The tips promote habit formation, nutrition awareness, avoidance of behavioural relapse, and reiterate guidance for pregnant women. Participants provided with a record-keeping logbook and access to an 'app' to self-monitor their weight and behaviours against the 10 target behaviours, during pregnancy and up to 6 weeks postpartum.
  Interventions: Behavioral: Healthy Habits in Pregnancy and Beyond
- Control group (No Intervention): The control group will receive 'usual' antenatal care which does not involve routinely delivered specific or standardised dietary advice.

INTERVENTIONS:
Behavioral: Healthy Habits in Pregnancy and Beyond — Habit-based intervention to support the development of 10 healthy dietary and activity behaviours for pregnant women with overweight or obesity.
  Other Names: Ten Top Tips for a Healthy Weight
  Arms: Healthy Habits in Pregnancy and Beyond intervention

SUMMARY:
More than 50% of pregnant women are considered to have a BMI that is classified as overweight or obese when they present for antenatal care. Overweight and obesity in pregnancy is associated with complications and poorer health outcomes for mothers and their babies, as well as risk for excessive gestational weight gain and postpartum weight retention, increasing the likelihood of long-term obesity for these women. There is also evidence that excess maternal weight and weight gain in pregnancy is associated with obesity in the offspring from early childhood through to adolescence. There is an urgent need for simple, effective interventions targeting lifestyle which can be delivered during routine healthcare.

The overall aim of this study is to pilot test the delivery of a brief, habit-based weight management intervention, 'Healthy Habits In Pregnancy and Beyond', for pregnant women with overweight and obesity (body mass index between 25.0 & <38.0 kg/m2) in early pregnancy, to gather preliminary information on the intervention and to establish the feasibility and acceptability of delivering this intervention into routine antenatal care and existing antenatal care pathways across four geographical locations in Northern Ireland and the Republic of Ireland.

This study is a two-arm randomised controlled feasibility study. Healthcare staff in four partner sites will be trained in introducing the study to the target sample and in delivering the intervention. 80 women will be recruited and randomised to control (n=40) or intervention group (n=40) (20 at each site). Women randomised to the intervention group will receive a brief intervention to encourage the development of ten healthy habits in relation to diet, physical activity and weight management, plus their local routine antenatal care. The intervention will be delivered by a designated midwife at each site or a member of the research team, and is aimed to be integrated into appointments already attended by women as part of routine antenatal care. Women randomised to the control group will receive their local routine antenatal care.

DETAILED DESCRIPTION:
The primary objective of the feasibility study is to provide a decision on whether to proceed to a full-scale, multicentre RCT.

The two-arm randomised controlled feasibility study will:

1. Assess the numbers of eligible pregnant women accessing the healthcare services at each partner healthcare site;
2. Assess screening, recruitment and attrition rates;
3. Assess willingness of healthcare staff to recruit women and deliver the HHIPBe intervention as part of routine antenatal clinical care;
4. Assess indicators of engagement with the intervention by women (self-reported logbooks/ app data/ qualitative post-intervention interviews);
5. Assess the acceptability of randomisation to a 'usual care' group and women's views on completion of study measures at each time-point;
6. Assess the acceptability of the intervention to women;
7. Assess fidelity of intervention implementation across each partner site i.e. was HHIPBe delivered as intended;
8. Trial the outcome measures that would be used in a full trial of HHIPBe (and gather data to inform a power calculation for a full trial) including assessment of: GWG, habit-formation and diet and activity behaviours up to 6 weeks postpartum; and health economics measures, alongside an exploration of the potential for data linkage to maternal and neonatal outcomes in each jurisdiction.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant Women.
* Body Mass Index between ≥25.0 kg/m2 and <38.0 kg/m2.
* Primiparous or Multiparous.
* Women capable of providing informed consent and of providing consent on behalf of their child.

Exclusion Criteria:

* Twin or multiple pregnancies.
* Insufficient English to understand intervention and written materials.
* Nutritional complications i.e. previous or current eating disorder, following a special diet, in receipt of specialist dietary advice.
* Pregnancy not viable as determined by the patient's clinical team.
* Have been referred to another weight management service by their clinical team during pregnancy that is not part of routine antenatal care.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-09-25 (Actual); Study Completion 2022-09-25 (Actual)

PRIMARY OUTCOMES:
Acceptability of the intervention | 6 weeks postpartum
  Interviews with participants and study-specific satisfaction rating scale (5 point scale from very satisfied to very dissatisfied)

SECONDARY OUTCOMES:
Feasibility of recruitment | During 4 month study recruitment period
  Number of women recruited to the study
Retention rate | End of study - 6 weeks postpartum
  Number of women completing the study
Acceptability to healthcare staff | Conducted during the 4 month study recruitment and 5 month intervention delivery periods
  Interviews with staff recruiting and delivering the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Michelle McKinley, PhD, Principal Investigator — Queen's University, Belfast
Locations (1):
- Centre for Public Health, Queen's University Belfast, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McClelland J, Gallagher D, Moore SE, McGirr C, Beeken RJ, Croker H, Eastwood KA, O'Neill RF, Woodside JV, McGowan L, McKinley MC. Development of a habit-based intervention to support healthy eating and physical activity behaviours for pregnant women with overweight or obesity: Healthy Habits in Pregnancy and Beyond (HHIPBe). BMC Pregnancy Childbirth. 2024 Nov 16;24(1):760. doi: 10.1186/s12884-024-06945-7. PMID 39550532